CLINICAL TRIAL: NCT05460286
Title: Comparing the Effects of Chiropractic Manipulation and Spinal Decompression Device Treatment on Lower Extremity Muscle Strength and Balance in Patients With Chronic Low Back Pain
Brief Title: Comparing the Effect of Chiropractic Manipulation and Spinal Decompression Device Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa AĞRAŞ (Other)
Responsible Party: Sponsor-Investigator, Mustafa AĞRAŞ, Principal Investigator, Bahçeşehir University
Organization: Bahçeşehir University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10466602
Record Dates: First submitted 2022-07-07; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Chronic Low-back Pain
Keywords: Balance; Chiropractic; Chronic low back pain; Muscle strength; Manipulation; Spinal decompression; Pain measurement; Range of motion; Recovery of function; Quality of life
MeSH Terms: interventions — Manipulation, Chiropractic

STUDY DESIGN:
Intervention Model Description: The individuals are randomly allocated into the CSMT or the SD groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSMT group (Experimental): Chiropractic Spinal Manipulative Treatment group
  Interventions: Other: Chiropractic Manipulation
- SD group (Experimental): Spinal Decompression group
  Interventions: Other: Spinal Decompression Device Treatment

INTERVENTIONS:
Other: Chiropractic Manipulation — 20 participants with low back pain existing more than 3 months was included in the CSMT group. Lumbar region chiropractic HVLA (High Velocity, Low Amplitude) spinal manipulation and/or sacroiliac joint chiropractic HVLA manipulation were applied to participants. Participants were treated three times with an interval of three days. Before and after treatment were evaluated lower extremity (hamstring and quadriceps) muscle strength with an isokinetic dynamometer (CSMI Humac-Norm), balance performance with BBS (Biodex Balance System), lumbar range of motion and mobility with inclinometer and hand finger floor distance (HFFD), low back pain intensity with visual analog scale (VAS), functional status with Modified Oswestry low back pain disability questionnaire (OSW), quality of life with Short form-36 (SF-36).
  Arms: CSMT group
Other: Spinal Decompression Device Treatment — 20 participants with low back pain existing more than 3 months was included in the SD group. Lumbar region spinal decompression (traction) device therapy was applied to participants, and as a standard of treatment was given a hot pack for 15 minutes before applying and a cold pack for 10 minutes after applying. Participants were treated three times with an interval of three days. Before and after treatment were evaluated lower extremity (hamstring and quadriceps) muscle strength with an isokinetic dynamometer (CSMI Humac-Norm), balance performance with BBS (Biodex Balance System), lumbar range of motion and mobility with inclinometer and hand finger floor distance (HFFD), low back pain intensity with visual analog scale (VAS), functional status with Modified Oswestry low back pain disability questionnaire (OSW), quality of life with Short form-36 (SF-36).
  Arms: SD group

SUMMARY:
This study is aimed to compare the effects of chiropractic spinal manipulative therapy and spinal decompression device treatment on lower extremity muscle strength, balance performance, lumbar range of motion and mobility, functional status, pain, and quality of life in patients with chronic low back pain.

After the approval of the ethics committee, the research was carried out in the physical therapy and rehabilitation clinic of Medipol Mega University Hospital. Individuals between the ages of 18-60, who had complaints of low back pain for the last three months and who voluntarily agreed to participate in the study were included in the study. 40 participants with low back pain existing more than 3 months were randomized into one of two groups as Chiropractic Spinal Manipulative Therapy (CSMT) and Spinal Decompression (SD). Lumbar region chiropractic HVLA (High Velocity, Low Amplitude) spinal manipulation and/or sacroiliac joint chiropractic HVLA manipulation was applied to CSMT group, and lumbar region spinal decompression (traction) device therapy was applied to SD group, and as a standard of treatment was given a hot pack for 15 minutes before applying and a cold pack for 10 minutes after applying. Both groups were treated three times with an interval of three days. Before and after treatment were evaluated lower extremity (hamstring and quadriceps) muscle strength with an isokinetic dynamometer (CSMI Humac-Norm), balance performance with BBS (Biodex Balance System), lumbar range of motion and mobility with inclinometer and hand finger floor distance (HFFD), low back pain intensity with visual analog scale (VAS), functional status with Modified Oswestry low back pain disability questionnaire (OSW), quality of life with Short form-36 (SF-36) in both groups. SPPS 25 (IBM Corp. Released 2017. IBM SPSS Statistics for Windows, Version 25.0. Armonk, NY: IBM Corp.) version was used to analyze the data.

DETAILED DESCRIPTION:
This study is aimed to compare the effects of chiropractic spinal manipulative therapy and spinal decompression device treatment on lower extremity muscle strength, balance performance, lumbar range of motion and mobility, functional status, pain, and quality of life in patients with chronic low back pain.

Chronic low back pain is a multifactorial disease that occurs especially in adults and has many negative effects on daily quality of life. This disease, which affects 70-80 percent of adults throughout their lives, creates significant limitation and high psycho-social burden in daily life due to the fact that the pain lasts more than 12 weeks. This leads to high health costs as well as loss of labor and economic burden.

The etiology of chronic low back pain varies according to the patient population, but the most common is mechanical and non-specific. 80-90 percent of low back pain is caused by mechanical low back pain, and 15-25 percent of these patients have chronic facet joint-induced low back pain caused by chronic inflammation and degeneration of the lumbar facet joints. Chronic low back pain is often thought to be caused by disc and/or vertebral degeneration, musculoskeletal sprain or strain, position of the spine, or movement-related disorders.

Limitation of movement increases due to pain and spasm seen in individuals with low back pain, and physical endurance decreases as a result of decreasing muscle strength and deteriorating posture due to non-use. As a result of this situation, the functional capacity and quality of life of individuals with low back pain are adversely affected.

In studies in individuals with low back pain, atrophy in multifidus and paraspinal muscles, delay in stimulation of the transversus abdominus muscle, decrease in hip abductor muscle strength and trigger points in the gluteus medius muscle have been shown. It has also been shown to have a decrease in hip extensor muscle strength, a decrease in hip flexion, and a significant decrease in hamstring muscle flexibility. In a study investigating knee extensor muscle strength, it was shown that the maximum voluntary contraction and isokinetic muscle strength of the knee extensors were reduced. It has been shown that individuals with chronic low back pain also have a weakened ability to balance due to decreased muscle strength, flexibility, endurance, and many physical changes.

Multifaceted treatment approaches are important because of the long-term and high cost of low back pain treatment. Medical treatment and conservative treatment (electrophysical agents, massage, traction, manipulation, exercise, etc.), public health and preventive rehabilitation programs constitute an important part of the treatment of low back pain.

Traction therapy is a broad term used to refer to any method of separation of the spine along its lower axis using mechanical force. It is used to reduce pain, especially in the cervical and lumbar regions. Traction therapy, which is one of the many treatments that mechanically drain the spine to treat chronic low back pain, has different types such as spinal traction, distraction, and non-surgical spinal decompression.

Spinal decompression (SD) therapy is a new method used as a conservative treatment for low back pain. Using movement and positioning with a traction table or similar motorized device is used to reduce pressure that can cause severe pain in the spine without any surgical procedure. Although it is generally suggested that this traction-based treatment is superior to existing classical traction devices, its basic principle is spinal distraction, which is thought to increase the distance between interververtebral discs by relaxing neural structures with its mechanical effects . Disc herniation or bulging creates a negative intervertebral pressure for the withdrawal and repositioning of disc material, and thanks to low pressure, it increases the fluid in the disc and the flow of fluids that nourish the disc.

Chiropractic consists of the Greek words chiro (hand) and practic (practice) and means "manual practice." Chiropractic, which is an evidence-based primary health care, is generally preferred by people with low back and neck pain in developed countries. In biomechanical disorders of the musculoskeletal and spinal systems that have not reached the surgical level, the complex of vertebral subluxation caused by isolated axis disorders, mechanical movement integrity and disruption of physiological functions or their negative effects on the nerve, muscle, ligaments, circulation and movement systems Chiropractic manipulations applied for the purpose of correction are an easy-to-apply, non-invasive, cost-effective and low form of treatment with side effects.

Although there are many studies in the literature in which the effects of conservative treatments used in the treatment of individuals with chronic low back pain are independently examined or compared with each other, there have been no studies comparing chiropractic manipulation and non-surgical spinal decompression treatments.

After the approval of the ethics committee, the research was carried out in the physical therapy and rehabilitation clinic of Medipol Mega University Hospital. Individuals between the ages of 18-60, who had complaints of low back pain for the last three months and who voluntarily agreed to participate in the study were included in the study. 40 participants with low back pain existing more than 3 months were randomized into one of two groups as Chiropractic Spinal Manipulative Therapy (CSMT) and Spinal Decompression (SD). Lumbar region chiropractic HVLA (High Velocity, Low Amplitude) spinal manipulation and/or sacroiliac joint chiropractic HVLA manipulation was applied to CSMT group, and lumbar region spinal decompression (traction) device therapy was applied to SD group, and as a standard of treatment was given a hot pack for 15 minutes before applying and a cold pack for 10 minutes after applying. Both groups were treated three times with an interval of three days. Before and after treatment were evaluated lower extremity (hamstring and quadriceps) muscle strength with an isokinetic dynamometer (CSMI Humac-Norm), balance performance with BBS (Biodex Balance System), lumbar range of motion and mobility with inclinometer and hand finger floor distance (HFFD), low back pain intensity with visual analog scale (VAS), functional status with Modified Oswestry low back pain disability questionnaire (OSW), quality of life with Short form-36 (SF-36) in both groups. SPPS 25 (IBM Corp. Released 2017. IBM SPSS Statistics for Windows, Version 25.0. Armonk, NY: IBM Corp.) version was used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain for more than 3 months
* Presence of sacroiliac and lumbar spine asymptomatic dysfunctions in tests

Exclusion Criteria:

* Not wanting to continue education
* Not being able to come to assessments
* Having low back pain after COVID-19
* Being spinal manipulation or spinal decompression treatment recently
* Having any neurological or psychiatric illness
* Having a fracture in the past
* Having a tumor in the past
* Lumbar disc hernias, spondylosis, spondylolisthesis
* Having a disease related to the cardiac and respiratory system
* Having an infectious, rheumatological, metabolic, and endocrine disease
* Having dislocation, osteoporosis, ankylosing spondylitis, discopathy, rheumatoid arthritis
* Having instability, acute myelopathy, or being anticoagulants treatments
* Having surgery recently

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Lower Extremity Muscle Strength: Hamstring and Quadriceps Isokinetic Test | 2 weeks
  In the measurement of lower extremity muscle strength of the participants, Quadriceps and Hamstring isokinetic peak torque values were measured with isokinetic dynamometer (CSMI-Cybex Humac-Norm Testing & Rehabilitation System). Maximal reciprocal concentric isokinetic knee extension and flexion of the participants were measured at three different angular speeds; slow (60°/s, 5 reps, 10 s rest), moderate (120°/s, 10 reps, 10 s rest) and fast (180°/s, 15 reps, 10 s rest)
Balance Performance: Postural Stability Test (PST), Fall Risk Test (FRT) and Balance Error Scoring System (BESS) | 2 weeks
  Static and dynamic balance performances of the participants were measured with the biodex balance system, which is a validated and reliable device that can be used to assess postural stability, balance error score and fall risk. This system, which can objectively measure balance performance, consists of a mobile platform, arm supports, screen and printer, whose surface can be tilted up to 20 degree in 360 degree range of motion. The platform can be adjusted as static or mobile (12 levels of movement amount; level 12 is the most stable, level 1 is the least stable level that can move up to 20 degree in each direction) according to the test to be applied.
Lumbal Region Range of Motion and Mobility Measurements: Inclinometer (Trunk Flexion and Extension) and Hand Finger-Floor Distance (HFFD) | 2 weeks
  Lumbal region range of motion of the participants (trunk flexion and extension) were measured with an inclinometer. The inclinometer, as its working principle, can be used in sagittal and frontal plane movements because it measures the angle between the in-app axis and the direction of gravity.
  Lumbar mobility of the participants was evaluated with the hand finger-floor distance (HFFD) test. Participants were leaned forward as much as they can, standing, hands-free, without bending their knees. The measurement of the distance between the third finger of the participants and the floor was recorded.
Pain Intensity Measurements: Visual Analog Scale (VAS-Rest and VAS-Movement) | 2 weeks
  Pain intensity measurements of the participants were evaluated with a visual analog scale (VAS-Rest and VAS-Movement) numbered equal intervals from 0 to 10 on a 10 cm line, which is used to digitize some values that cannot be measured numerically. 0 means no pain and 10 means unbearable pain. Thus, participants was asked to mark the intensity of pain they perceive.
Functional Status Measurement: Oswestry Low Back Pain Disability Questionnaire (OSW) | 2 weeks
  Functional status measurement of the participants were evaluated with a Oswestry Low Back Pain Disability Questionnaire (OSW). This questionnaire measures disability in 10 different aspects (intensity of pain, personal care, lifting, walking, sitting, standing, sleep, social life, travel, change in the amount of pain) in order to evaluate the effect of low back pain on activities of daily living. Each item consists of six options in itself. The patient marks the option that best expresses his or her condition. The first option gets a score of "0" and the sixth option gets a score of "5". The level of functionality expressed by the scores is as follows; (0-4 points no disability), (5-14 points mild), (15-24 points moderate), (25-34 points severe), (35-50 points range of complete functional disability). The minimum score obtained from the scale is 0, and the maximum score is 50. 50 points indicate that functional disability is at the highest level.
Quality of Life Measurements: Short-Form 36 (SF-36) | 2 weeks
  Quality of life measurement of the participants were evaluated with a Short Form-36, which is the most commonly used quality of life scale in the medical field. This questionnaire consists of 8 sub-scales with a total of 36 items that evaluate physical and mental health. These subscales are physical function, physical role limitation, pain, general health, vitality, social function, emotional role limitation, and mental health. It was found to be valid and reliable in patients with osteoarthritis and chronic low back pain. The scores range from 0-100, with 100 points indicating the best health condition and 0 points the worst health condition.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Veysel ÖZDEN, PhD., Study Director — Bahçeşehir University; Sena TOLU, Assoc. Prof., Study Director — Medipol University; Mustafa AĞRAŞ, MSc., Principal Investigator — Bahçeşehir University
Locations (1):
- Medipol Mega University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson GB. Epidemiological features of chronic low-back pain. Lancet. 1999 Aug 14;354(9178):581-5. doi: 10.1016/S0140-6736(99)01312-4. PMID 10470716
- [Background] Parthan A, Evans CJ, Le K. Chronic low back pain: epidemiology, economic burden and patient-reported outcomes in the USA. Expert Rev Pharmacoecon Outcomes Res. 2006 Jun;6(3):359-69. doi: 10.1586/14737167.6.3.359. PMID 20528528
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] Manusov EG. Evaluation and diagnosis of low back pain. Prim Care. 2012 Sep;39(3):471-9. doi: 10.1016/j.pop.2012.06.003. PMID 22958556
- [Background] Prather H, Cheng A, Steger-May K, Maheshwari V, Van Dillen L. Hip and Lumbar Spine Physical Examination Findings in People Presenting With Low Back Pain, With or Without Lower Extremity Pain. J Orthop Sports Phys Ther. 2017 Mar;47(3):163-172. doi: 10.2519/jospt.2017.6567. Epub 2017 Feb 3. PMID 28158964
- [Background] Sadler S, Cassidy S, Peterson B, Spink M, Chuter V. Gluteus medius muscle function in people with and without low back pain: a systematic review. BMC Musculoskelet Disord. 2019 Oct 22;20(1):463. doi: 10.1186/s12891-019-2833-4. PMID 31638962
- [Background] Peterson CK, Bolton J, Humphreys BK. Predictors of improvement in patients with acute and chronic low back pain undergoing chiropractic treatment. J Manipulative Physiol Ther. 2012 Sep;35(7):525-33. doi: 10.1016/j.jmpt.2012.06.003. Epub 2012 Jul 31. PMID 22858233
- [Background] de Sousa CS, de Jesus FLA, Machado MB, Ferreira G, Ayres IGT, de Aquino LM, Fukuda TY, Gomes-Neto M. Lower limb muscle strength in patients with low back pain: a systematic review and meta-analysis. J Musculoskelet Neuronal Interact. 2019 Mar 1;19(1):69-78. PMID 30839305
- [Background] Fasuyi FO, Fabunmi AA, Adegoke BOA. Hamstring muscle length and pelvic tilt range among individuals with and without low back pain. J Bodyw Mov Ther. 2017 Apr;21(2):246-250. doi: 10.1016/j.jbmt.2016.06.002. Epub 2016 Jun 16. PMID 28532865
- [Background] da Silva RA, Vieira ER, Fernandes KBP, Andraus RA, Oliveira MR, Sturion LA, Calderon MG. People with chronic low back pain have poorer balance than controls in challenging tasks. Disabil Rehabil. 2018 Jun;40(11):1294-1300. doi: 10.1080/09638288.2017.1294627. Epub 2017 Mar 10. PMID 28282992